CLINICAL TRIAL: NCT04454255
Title: Evaluating the Educational Benefits of Tablet-based Serious Games to Promote Speech Production in Instrumented Young Children With Hearing Disabilities
Brief Title: Benefits of Tablet-based Serious Games to Promote Speech Production in Young Children With Hearing Disabilities
Acronym: FunSpeech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Angelica Perez Fornos, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ID 2019-02138
Record Dates: First submitted 2020-03-05; First posted 2020-07-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Deafness; Hearing Loss
Keywords: Serious game; Speech development; Speech production; Cochlear implant; Hearing aid; Bone anchored hearing aid
MeSH Terms: conditions — Deafness; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Cross-over, repeated-measures, open without masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primo-FunSpeech (Experimental): Participants will begin the study by a period using FunSpeech (45 days) followed by a control period without the game (45 days). This sequence will be repeated once.
  Interventions: Behavioral: FunSpeech
- Primo-control (Experimental): Participants will begin the study by a control period without the game (45 days) followed by a period using FunSpeech (45 days). This sequence will be repeated once.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: FunSpeech — Weekly sessions of regular speech therapy as regularly performed for the individual participant (one hour, once or twice a week) and parent-supervised home use of a serious game. It will be recommended to use FunSpeech every day, 15 minutes per day.
  Arms: Primo-FunSpeech
Behavioral: Control — Weekly sessions of regular speech therapy as regularly performed for the individual participant (one hour, once or twice a week).
  Arms: Primo-control

SUMMARY:
Learning to speak is a major challenge for children with hearing impairments. Nowadays, special devices such as conventional hearing aids, bone-anchored hearing aids (BAHA) or cochlear implants (CI) allow successful rehabilitation of patients with hearing disabilities. To obtain maximum benefit from these technical aids, instrumented hearing impaired children require specific and intensive speech therapy to compensate for speech development delays. In addition, it is also of primary importance that during daily life (e.g., at home, at school) children are provided with sufficient and good quality auditory stimulation.

The main goal of this project is to encourage speech production with an edutainment tool that can be used at home and that is adapted to the specific needs of young hearing impaired children. For this purpose, the investigators have recently designed an innovative educational solution: FunSpeech, a tablet-based set of video games that respond exclusively to sound and speech. The aim of this serious game is to encourage hearing impaired children to produce controlled sounds in terms of rhythm, intensity, and pitch. These are the main abilities required for controlled speech production. Finally, this serious game aims to support the parents' key role in the speech learning process by offering an effective solution that is easy to use at home with young children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild to profound hearing loss,
* Optimum instrumented hearing (hearing aids, BAHA or CI),
* Language development delay confirmed by a speech therapist,
* Enough sensorimotor, cognitive and communication skills to play with tablet-based games,
* French mother tongue

Exclusion Criteria:

* Additional impairments which affect language development or the use of FunSpeech (e.g. motor, orofacial, sensory, cognitive),
* Refusal of the participant's representative(s) to participate in the study,
* Refusal of the participant's representative(s) to participate in a modality of the study,
* If the child/participant refuses to collaborate in two measures of language level.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Parental inventory (questionnaire) and observation grid of speech production skills completed by the speech therapist. | 6 months
  Quantitative and qualitative assessments of spoken language level.

SECONDARY OUTCOMES:
Game usage (total play time, frequency of play sessions, list of games used, gameplay goals achieved) | 6 months
  This data will be gathered via a tracking system implemented in the game and parental interviews (questionnaires).

OTHER OUTCOMES:
Ergonomy questionnaire (ease of use) on a seven-point Likert scale (1 = strongly disagree to 7 = strongly agree). | 6 months
  Game usability
Open interview (issues/concerns about the game) | 6 months
  Acceptance degree of the game

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No